CLINICAL TRIAL: NCT03733093
Title: PREVAIL VIII: A CoHOrt Clinical, Viral, and ImmuNOlogic Monitoring Study of People Living With Retroviral Infection in Liberia (HONOR)
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999919014; 19-I-N014
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01-08

CONDITIONS: HIV
Keywords: HIV; Opportunistic Diseases; Tuberculosis; AIDS; Sexually Transmitted Infection; Natural History
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: HIV Positive

SUMMARY:
Background:

There are many people living with human immunodeficiency virus (HIV) infection in Liberia. Most experts consider HIV an epidemic there. Researchers want to collect health data from Liberians with HIV over several years. This may help HIV prevention and treatment programs in Liberia.

Objective:

To learn more about how HIV affects people in Liberia.

Eligibility:

People with HIV in Liberia

Design:

Participants will be screened with a blood sample.

Participants will visit the study clinic about 10 times over 3 years. They will need to return to the clinic after some visits to get test results. The visits will be closer together during the first part of the study and less frequent later.

At each study visit, participants will:

* Have a brief physical exam
* Answer questions about how they are feeling and what medicines they are taking
* Have blood taken from an arm vein by a needle
* Give urine samples

Participants ages 12 years or older may be asked questions about HIV risk behaviors. These include sex practices and drug use. Participants ages 18 years or older may be asked how their

HIV infection makes them feel emotionally.

Participants may be asked to join a research substudy. This will be about tuberculosis (TB) testing in people with HIV. For this substudy, participants will have a TB skin test. A small amount of liquid will be injected under the skin on the arm.

Participants will return to the clinic a few days later. The test area will be checked. They will get their test results.

DETAILED DESCRIPTION:
Resources for management of HIV-positive individuals are extremely limited in the West African country of Liberia, and many knowledge gaps exist about the nature of the HIV epidemic in this country. While the prevalence is likely low compared to other regions in Sub-Saharan Africa, the burden of disease is likely high given the current state of the Liberian health care system, despite attempts to improve HIV treatment services and coverage. The Ebola epidemic of 2014-2016 created tremendous strain on a health care system already weakened by years of civil strife, and it is suspected that care for many HIV-positive individuals was disrupted by this event. Currently, clinicians do not have regular access to measurements of CD4 levels or viral loads, making management of people living with HIV in Liberia difficult. While there is some access to antiretroviral (ARV) medications through the National AIDS and Sexually Transmitted Infection (STI) Control Program, several details, including the extent of this access and the impact on disease outcomes, remain unknown. This cohort study will examine these basic factors; attempt to characterize major social/demographic, clinical, immunologic, and virologic features of HIV/AIDS; and investigate the course of HIV disease, including rates of hospitalization, frequencies of ARV regimen modifications, and incidence of certain opportunistic diseases, STIs, other co-infections, and non-AIDS comorbidities among those who are enrolled. Study participants will attend periodic study visits over 3 years. Clinical information will be collected, as will blood and urine samples for clinical and research tests. This protocol is not designed to estimate the prevalence of HIV infection; however, it provides a unique opportunity to generate quality data to understand the course and epidemiology of HIV and AIDS in Liberia. It also provides an opportunity to contribute to the quality and impact of HIV prevention, treatment, and care programs in Liberia.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals of any age and gender must meet all of the following criteria to be eligible for study participation:

1. HIV infection confirmed by HIV-1/2 enzyme-linked immunosorbent assay (ELISA) and confirmatory test or positive assay for HIV-1 pVL.
2. Ability to provide informed consent.
3. Willingness to allow storage of biological samples for research testing.
4. Willingness to be followed by a participant tracker.

EXCLUSION CRITERIA:

Individuals meeting the following criterion will be excluded from study participation:

1. Any condition that, in the opinion of the investigator, would compromise the safety of the study subject or staff, or would prevent proper conduct of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cohort of individuals currently receiving or initiating care for HIV infection in Margibi and Montserrado Counties, Liberia.
Sampling Method: Non-Probability Sample
Enrollment: 1377 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Description of disease course | Months 1,3,6,12,18,24,30,36
  Description of the course of HIV disease in the study population as a whole or by subgroup.
Characteritics of study population | Baseline
  Description of major social/demographic, clinical, immunologic, and virologic characteristics of HIV disease in the study population at baseline.

SECONDARY OUTCOMES:
ARV Genotypic Resistance Mutations | 1 year
  Determine ARV genotypic resistance mutations within 1 year of study initiation on stored samples from a subset of participants with HIV-1 pVL >1000 copies/mL at baseline (+/- ART) or at other early study timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Migueles, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (4):
- Liberia (4):
  - C.H. Rennie Hospital, Kakata
  - John F. Kennedy (JFK) Medical Center, Monrovia
  - Redemption Hospital, Monrovia
  - Duport Road Clinic, Paynesville

IPD SHARING:
Plan to Share IPD: No
De-identified data will be shared